CLINICAL TRIAL: NCT03531931
Title: Single-arm Exploratory Clinical Study on the Second-line Treatment of Advanced Gastric Cancer With Apatinib Mesylate Plus Capecitabine
Brief Title: Apatinib Combined With Capecitabine Second-line Treatment of Advanced Gastric Cancer: a Single-arm Exploratory Clinical Pilot Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: 20180509
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Progression-free Survival;Progression-free Survival;Disease Control Rate; Safety
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Apatinib/Capecitatine — Apatinib is a tyrosine kinase inhibitor that selectively inhibits the vascular endothelial growth factor receptor-2 (VEGFR2), now being developed by Jiangsu Hengrui Medicine (China). Even at a low concentration apatinib can still perform magnificent VEGFR2 inhibitory activities, meanwhile at little higher concentration it can inhibit PDGFR and kinases as well, such as c-Kit and c-Src .The action sites of apatinib are the intracellular ATP binding site of the protein tyrosine receptor. Pharmacodynamical study shows that apatinib is able to inhibit the tyrosine kinase activity of VEGFR, block signal conduction after the combination of VEGF, finally contribute to stopping new blood vessel formation in tumor tissue.

SUMMARY:
Gastric cancer is the one of the leading cause of cancer death in the worldwide. Gastric cancer originates from the most superficial mucosal epithelial cells of the stomach wall, which can occur in various parts of the stomach, and can invade different depths and breadth of the gastric wall. Without chemotherapy treatment the GC patients' Median Survival Time (MST) lasts only 3-4 months. Although treated with multi-chemotherapy MST has been improved, the drugs show strong toxicities in the patients. Thus the more accurate, lower toxicity, targeted antitumor drugs are put into second-line treatment program for advanced gastric cancer.

Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with GC. The purpose of this study is to determine whether apatinib plus capecitatine can improve progression free survival in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age：18~75 years; 2. Subjects with pathologically (included histologically or cytologically) confirmed gastric adenocarcinoma, unresectable local advanced or metastatic tumors; 3. Only second-line gastric cancer patients in late phase and at least one month interval from the latest chemotherapy treatment; 4. Previous treatment program without apatinib or capecitabine or any other antiangiogenic medications; 5. Subjects with at least one measurable lesion (defined by RECIST ,version 1.1), which is confirmed by computed tomography (CT) scan or MRI≥10mm .

  6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 7. Survival expectation≥ 3 months; 8. Subjects were recovered from damages caused by other treatments, with the interval ≥ 6 weeks for the treatment of the Nitro or Mitomycin, and 4 weeks for other cytotoxic drugs, radiotherapy or surgery, and the wound is completely healed 9. Subjects without severe heart, lung or liver dysfunction, no jaundice and digestive tract obstruction, and acute infection associated 10. The main organs function normally, and meet the following standards:
  1. Standard of blood routine examination conforms to ( no blood transfusion within 14 days):

     1. Hemoglobin (HB)≥ 80 g/L;
     2. Leukocyte(WBC)≥3.5×109/L;
     3. Absolute neutrophil count (ANC)≥1.5×109/L;

     c. Platelet count (PLT) ≥75×109/L；
  2. Sufficient liver function:

     1. Bilirubin(BIL) <1.25×the upper limit of normal (ULN);
     2. Alanine aminotransferase (ALT), and Aspartate aminotransferase (AST) <2.5×(ULN), Glutamic-pyruvic transaminase(GPT)≤1.5×ULN. If liver metastases occur, ALT and AST <5×(ULN), GPT≤3×(ULT);
     3. Serum Creatinine(Cr) ≤1.0×（ULN）, or creatinine clearance > 50 mL/min( calculated per the Cockcroft and Gault formula); 11. Females of childbearing potential must receive a pregnancy test within 7 days before participating ( including serum), and the results are negative, and also willingly take appropriate methods for contraception during the trial or within 8 weeks after the latest medication. Males should be surgically sterilized or agreed to use the appropriate contraceptive method during the trial or within 8 weeks after the latest medication.

        12. Subjects provided written informed consent before participating, willing and able to comply with all aspects of the protocol.

        Exclusion Criteria:
* 1. Pregnant or lactating females; 2. Subjects previously or meanwhile with other malignancies, except cured cutaneous basal cell carcinoma and cervical carcinoma; 3. Subjects with severe heart, liver, kidney disease; with uncontrolled symptomatic brain metastases; with neurological and psychiatric disorders; with severe infection; 4. With high blood pressure and treated with antihypertensive drugs still unable to reduce to the normal range (systolic pressure > 140 mmhg, diastolic pressure >90 mmhg ); 5. With level I above coronary heart disease, arrhythmia (including QTc period extended, male >450 ms, female >470 ms) and cardiac insufficiency; 6. with obvious gastrointestinal bleeding tendencies, include the following situation: locally active ulcer lesions, fecal occult blood (+ +), and within 2 months with a history of black stool or vomiting of blood; coagulation dysfunction (INR>1.5, APTT>1.5 ULN); 7. With Previous history of cardio-cerebral vascular disease, now still take oral thrombolytic drugs or anticoagulant drugs; 8. Urine protein examination confirmed positive (urine protein detection ++ or above, or 24-hour urine protein quantitative detection >1.0g); 9. According to the investigators' judgment, subjects who put other subjects at risk of the safety or disturb their clinical trial devolpment; 10. There are factors that affect oral administration (such as inability to swallow, persistent uncontrolled nausea, vomiting, chronic diarrhea, and intestinal obstruction); 11. Subjects confirmed unsuitable for the clinical trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with pathologically (included histologically or cytologically) confirmed gastric adenocarcinoma, unresectable local advanced or metastatic tumors; Only second-line gastric cancer patients in late phase and at least one month interval from the latest chemotherapy treatment;
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 month
  To assess progression-free survival (PFS) in subjects treated with apanitib plus capecitatine as a second-line treatment in whom with advanced gastric cancer or adenocarcinoma of the stomach-esophagus joint.

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No